CLINICAL TRIAL: NCT02875054
Title: Camp High 5 2016: Evaluation of the Effect on Upper Limb Function
Brief Title: Camp High 5: Evaluation of the Effect on Upper Limb Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 16-00990
Record Dates: First submitted 2016-08-12; First posted 2016-08-23 (Estimated); Last update posted 2017-04-21 (Actual); Status verified 2017-04

CONDITIONS: Neurological Injury; Hemiplegia
MeSH Terms: conditions — Trauma, Nervous System; Hemiplegia | interventions — Constraint Induced Movement Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Continued Casting (Active Comparator): Participants with 24 hour cast wear (continued casting) for the entire duration of the constraint portion of camp (2 initial weeks).
  Interventions: Behavioral: Constraint induced movement therapy (CIMT); Behavioral: Hand-arm bimanual intensive training (HABIT)
- Intermittent Casting (Active Comparator): Participants who wear a univalve cast for 3 hours of constraint camp with home exercise program of 2 hours cast wear on the weekends (intermittent casting).
  Interventions: Behavioral: Constraint induced movement therapy (CIMT); Behavioral: Hand-arm bimanual intensive training (HABIT)

INTERVENTIONS:
Behavioral: Constraint induced movement therapy (CIMT) — Involves forcing use of ones affected upper extremity (UE) by physically restraining the less affected upper extremity
Behavioral: Hand-arm bimanual intensive training (HABIT) — Facilitates the translation of gains to improve goal-directed bimanual performance.

SUMMARY:
Randomized control trial to evaluate uni-manual and bimanual upper limb function as well as compare outcomes of varied cast wear in children with hemiplegic cerebral palsy (CP) following a hybrid camp model of modified constraint induced movement therapy (mCIMT) and hand-arm bimanual intensive training (HABIT).

ELIGIBILITY:
Inclusion Criteria:

* Participants will range from 2 years to 11 years 11 months of age at time of enrollment. Children under 5 years of age will attend a morning session and children 6 years and older will attend an -Diagnosis: hemiplegia resulting from a neurological Injury
* Manual Ability Classification System or Mini Manual Ability Classification System classification I-III

Exclusion Criteria:

* Botox injection within past 6 months or planned for within 6 months post camp
* Inability to follow commands
* Family unable to commit to daily sessions for 4 weeks
* Unable to tolerate assigned casting protocol (3-24 hours) daily for 4 weeks

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2017-01-01 (Actual); Study Completion 2017-01-01 (Actual)

PRIMARY OUTCOMES:
Pediatric Motor Activity Log | 6 Months
  parent questionnaire to determine how well and how often the family perceives the child Spontaneously uses their affected Upper Extremity throughout the day at home. This assessment is scored by adding up the parental score and getting an average score.
Assisting Hand Assessment | 6 Months
  Test of hand function in children with difficulties using one of their hands. The AHA measures how effectively the affected hand and arm is used in bimanual performance.
Melbourne-2 | 6 Months
  Test of unilateral upper limb function is a validated and reliable tool for evaluating quality of upper limb movement in children with neurological conditions aged 2.5 to 15 years.

CONTACTS AND LOCATIONS:
Overall Officials: Renat Sukhov, MD, Principal Investigator — New York University Medical School
Locations (1):
- New York University School of Medicine, New York, New York, United States